CLINICAL TRIAL: NCT04245735
Title: The Role of Peripheral Perfusion Index in Evaluating the Success of Peripheral Nerve Block in Children Under Sedation
Brief Title: The Role of Perfusion Index in Children
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Erzincan University (Other)
Collaborators: Derince Training and Research Hospital (Other)
Responsible Party: Principal Investigator, İLKE KÜPELİ, assoc. prof., Derince Training and Research Hospital
Other Study IDs: EBYU PNB CHILDREN
Record Dates: First submitted 2020-01-26; First posted 2020-01-29 (Actual); Last update posted 2020-12-01 (Actual); Status verified 2020-11

CONDITIONS: Perfusion Index
MeSH Terms: interventions — Perfusion Index

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Diagnostic Test: perfusion index — To test the objective role of perfusion index in assessing the success of the peripheral nerve block in children under sedation.

SUMMARY:
The purpose of our study is to test the usability of the perfusion index in evaluating the success of the peripheral nerve block applied under sedation in children.

ELIGIBILITY:
Inclusion Criteria:

* will undergo elective upper limb surgery,
* 2- 10 years old,
* ASA I

Exclusion Criteria:

* have regional anesthesia contraindications,
* allergic to local anesthetics,
* having an infection at the injection site
* patients who do not accept the procedure

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 60 patients with ASA 1 between the ages 2-10 who will undergo elective upper extremity surgery will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2021-08-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
perfusion index | 6 months
  To test the objective role of perfusion index in assessing the success of the peripheral nerve block in children under sedation.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Abdelnasser A, Abdelhamid B, Elsonbaty A, Hasanin A, Rady A. Predicting successful supraclavicular brachial plexus block using pulse oximeter perfusion index. Br J Anaesth. 2017 Aug 1;119(2):276-280. doi: 10.1093/bja/aex166. PMID 28854539
- [Result] Kus A, Gurkan Y, Gormus SK, Solak M, Toker K. Usefulness of perfusion index to detect the effect of brachial plexus block. J Clin Monit Comput. 2013 Jun;27(3):325-8. doi: 10.1007/s10877-013-9439-4. Epub 2013 Feb 10. PMID 23397432
- [Result] Galvin EM, Niehof S, Verbrugge SJ, Maissan I, Jahn A, Klein J, van Bommel J. Peripheral flow index is a reliable and early indicator of regional block success. Anesth Analg. 2006 Jul;103(1):239-43, table of contents. doi: 10.1213/01.ane.0000220947.02689.9f. PMID 16790660
- [Result] Sebastiani A, Philippi L, Boehme S, Closhen D, Schmidtmann I, Scherhag A, Markstaller K, Engelhard K, Pestel G. Perfusion index and plethysmographic variability index in patients with interscalene nerve catheters. Can J Anaesth. 2012 Dec;59(12):1095-101. doi: 10.1007/s12630-012-9796-3. Epub 2012 Oct 2. PMID 23055034
- [Result] Xu Z, Zhang J, Shen H, Zheng J. Assessment of pulse oximeter perfusion index in pediatric caudal block under basal ketamine anesthesia. ScientificWorldJournal. 2013 Sep 19;2013:183493. doi: 10.1155/2013/183493. eCollection 2013. PMID 24174910